CLINICAL TRIAL: NCT05789355
Title: Effect of NUV001 Supplementation for 120 Days in Patients Suffering From Sickle Cell Disease (SCD) S Homozygous (SS) Genotype: A Pilot Study
Brief Title: Effect of NUV001 Supplementation in Patients Suffering From Sickle Cell Disease (SCD)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: LGD (Industry)
Collaborators: CEN Biotech (Industry); Assistance Publique Hopitaux De Marseille (Other); Etablissement Français du Sang (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Safety-DRNUV001- SCD
Record Dates: First submitted 2023-02-28; First posted 2023-03-29 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Sickle Cell Disease
Keywords: safety; tolerance; SS genotype of sickle cell disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Intervention Model Description: Single-center, prospective, open-label pilot study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NUV001 (Experimental): Daily supplementation with NUV001 1000 mg
  Interventions: Dietary Supplement: NUV001

INTERVENTIONS:
Dietary Supplement: NUV001 — Daily supplementation with NUV001 at 1000 mg (4 tablets of 250 mg each) for 90 days with a prolonged follow-up of 1 month (30 days) after stopping the supplementation

SUMMARY:
This is a pilot study of daily dosing of NUV001 as a dietary supplement in 12 sickle cell disease patients with 3 months of follow-up plus 1 month after supplementation.The present study is designed to evaluate, first, the safety and tolerability parameters as well as to measure the plasma and urinary residues of daily oral doses of NUV001. Secondly, the study will evaluate the impact of NUV001 on biological parameters and quality of life of patients.

DETAILED DESCRIPTION:
This is a monocentric, prospective, open label pilot study designed for 12 adult patients suffering of Sickle Cell disease (SCD) SS genotype each 12 receiving the active supplementation of NUV001, 1000mg/day (4 x 250 mg tablet) for 3 months of follow-up plus 1 month after supplementation. A stratification according to the medical treatment is planned. At least 2 patients suffering of SCD SS genotype without hydroxyurea treatment and maximum 10 patients suffering of SCD SS genotype in association with hydroxyurea treatment. If a subject is withdrawn from this study part, the subject may be replaced as necessary with another subject assigned to the same treatment at the discretion of the sponsor's team in consultation with the investigator.

The current study is designed to assess in the first part, the safety, tolerability, plasma, and urine residual rate parameters of daily oral doses of NUV001 as dietary supplement n adult patients suffering of sickle cell disease SS genotype. In a second part, the study will assess the pharmacological impact of NUV001 on biological parameters and the quality of life in patient suffering of sickle cell disease SS genotype.

ELIGIBILITY:
Inclusion Criteria:

1. Man or woman comprised between 18 and 60 years old.
2. Patients diagnosed with homozygous sickle cell anemia of SS genotype (documented by genotyping).
3. Females of childbearing potential should be using one of the following acceptable methods of birth control:

   * Intrauterine Device (IUD) in place for at least 60 days prior to the first dose of the study throughout the study and for 30 days after completion of the study.
   * Hormonal contraceptives for at least 90 days prior to the first dose of the study throughout the study, and for 30 days after study completion.
4. Patients whose weight is greater than 50 kg.
5. Patient that has been treated with an anti-sickling agent (Hydroxyurea) within six months of the screening visit, must maintain the therapy continuous and unmodified for at least six months with the intent to continue for the duration of the study.
6. Patient available to attend on an outpatient basis for visits provided for in the protocol and able to complete the data collection documents (and quality of life scale).
7. Patient has given written informed consent.
8. Patient with health insurance scheme

Exclusion Criteria:

1. Patient with known or suspected allergy to any ingredient of the food supplement .
2. Patient having consumed food supplements containing tryptophan, glutamine or vitamin B3 in its various forms (nicotinic acid/niacin and nicotinamide) during the month before selection
3. Patient has a significant medical condition that required hospitalization (other than sickle cell crisis) within two months of the screening visit.
4. Patient has serum albumin < 3.0 g/dl.
5. Patient has been transfused and received any blood products within three months of the Screening Visit.
6. Patient has been hospitalized for acute vaso-occlusive crisis within one months of the Screening Visit.
7. Patient has clinically significant, cardiovascular or liver disease, renal or lung insufficiency or lymphopenia (with clinically significant abnormal results on the screening bioassays: complete blood count, transaminases (ASAT, ALAT, GGT, ALP), bilirubin, creatinine, CPK, Ionogram, blood glucose, lipid profile).
8. Patients with diagnosed cancer in the past 2 years
9. Pregnant or lactating woman. Woman of childbearing potential should have a negative (serum or urinary TBD) pregnancy test at screening and a negative urine pregnancy test at inclusion prior to administration of the Study Product.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | between Day 0 and Day 30
  Subject incidence of treatment-emergent Adverse events (AEs) and Severe adverse events. Including Hospitalization days and Vaso-occlusive crisis occurrences.
Incidence of treatment-emergent adverse events | between Day 0 and Day 60
  Subject incidence of treatment-emergent Adverse events (AEs) and Severe adverse events. Including Hospitalization days and Vaso-occlusive crisis occurrences.
Incidence of treatment-emergent adverse events | between Day 0 and Day 90
  Subject incidence of treatment-emergent Adverse events (AEs) and Severe adverse events. Including Hospitalization days and Vaso-occlusive crisis occurrences.
Incidence of treatment-emergent adverse events | between Day 0 and Day 120
  Subject incidence of treatment-emergent Adverse events (AEs) and Severe adverse events. Including Hospitalization days and Vaso-occlusive crisis occurrences.
Incidence of treatment-emergent clinically significant changes in clinical laboratory safety tests | between Day 0 and Day 30
  Subject incidence of treatment-emergent clinically significant changes in clinical laboratory safety tests (Blood formulation, Inflammation parameters, Conjugated and free Bilirubin, alanine and aspartate aminotransferases (ASAT, ALAT),gamma-glutamyltransferase (GGT) and alkaline phosphatase (ALP), Creatine phosphokinase (CPK), Creatine, Urea, Creatinuria, Proteinuria, creatinine clearance)Ionogram Na/K/Cl, fasting blood glucose, albumine)
Incidence of treatment-emergent clinically significant changes in clinical laboratory safety tests | between Day 0 and Day 60
  Subject incidence of treatment-emergent clinically significant changes in clinical laboratory safety tests (Blood formulation, Inflammation parameters, Conjugated and free Bilirubin, alanine and aspartate aminotransferases (ASAT, ALAT),gamma-glutamyltransferase (GGT) and alkaline phosphatase (ALP), Creatine phosphokinase (CPK), Creatine, Urea, Creatinuria, Proteinuria, creatinine clearance)Ionogram Na/K/Cl, fasting blood glucose, albumine)
Incidence of treatment-emergent clinically significant changes in clinical laboratory safety tests | between Day 0 and Day 90
  Subject incidence of treatment-emergent clinically significant changes in clinical laboratory safety tests (Blood formulation, Inflammation parameters, Conjugated and free Bilirubin, alanine and aspartate aminotransferases (ASAT, ALAT),gamma-glutamyltransferase (GGT) and alkaline phosphatase (ALP), Creatine phosphokinase (CPK), Creatine, Urea, Creatinuria, Proteinuria, creatinine clearance)Ionogram Na/K/Cl, fasting blood glucose, albumine)
Incidence of treatment-emergent clinically significant changes in clinical laboratory safety tests | between Day 0 and Day 120
  Subject incidence of treatment-emergent clinically significant changes in clinical laboratory safety tests (Blood formulation, Inflammation parameters, Conjugated and free Bilirubin, alanine and aspartate aminotransferases (ASAT, ALAT),gamma-glutamyltransferase (GGT) and alkaline phosphatase (ALP), Creatine phosphokinase (CPK), Creatine, Urea, Creatinuria, Proteinuria, creatinine clearance)Ionogram Na/K/Cl, fasting blood glucose, albumine)
Incidence of treatment-emergent clinically significant changes in Vital Signs | between Day 0 and Day 30
  Subject incidence of treatment-emergent clinically significant changes in vital signs (systolic and diastolic blood Pressure, Pulse Rate and Body temperature)
Incidence of treatment-emergent clinically significant changes in Vital Signs | between Day 0 and Day 60
  Subject incidence of treatment-emergent clinically significant changes in vital signs (systolic and diastolic blood Pressure, Pulse Rate and Body temperature)
Incidence of treatment-emergent clinically significant changes in Vital Signs | between Day 0 and Day 90
  Subject incidence of treatment-emergent clinically significant changes in vital signs (systolic and diastolic blood Pressure, Pulse Rate and Body temperature)
Incidence of treatment-emergent clinically significant changes in Vital Signs | between Day 0 and Day 120
  Subject incidence of treatment-emergent clinically significant changes in vital signs (systolic and diastolic blood Pressure, Pulse Rate and Body temperature)

SECONDARY OUTCOMES:
Change in Lactate dehydrogenase (LDH) levels | Day 0, Day 15, Day 30, Day 60, Day 90, Day 120.
  Lactate dehydrogenase (LDH) levels evolutions from baseline
Change in Hemoglobin (HGB) levels | Day 0, Day 15, Day 30, Day 60, Day 90, Day 120.
  Hemoglobin (HGB) levels evolutions from baseline.
Change in Hematocrit (HCT) | Day 0, Day 15, Day 30, Day 60, Day 90, Day 120.
  Hematocrit (HCT) evolutions from baseline.
Change in circulating level of red line cell precursors | Day 0, Day 15, Day 30, Day 60, Day 90, Day 120.
  circulating level of red line cell precursors (basophilic, polychromic and orthochromatic / reticulocytes erythroid cells) evolutions from baseline measured by flow cytometry
Change in mean corpuscular volume (MCV) | Day 0, Day 15, Day 30, Day 60, Day 90, Day 120.
  mean corpuscular volume (MCV) evolutions from baseline measured
Change in mean corpuscular hemoglobin content (MCHT) | Day 0, Day 15, Day 30, Day 60, Day 90, Day 120.
  mean corpuscular hemoglobin content (MCHT) evolutions from baseline measured
Change in reticulocyte level | Day 0, Day 15, Day 30, Day 60, Day 90, Day 120.
  reticulocytes count expressed in percentage of red blood cells
F-Hemoglobin | Day 0, Day 15, Day 30, Day 60, Day 90, Day 120.
  F-Hemoglobin (HbF) level, % of F-cells, Distribution of HbF within F-cells (% of high and low F-cells) evolutions from baseline.
Circulating irreversibly sickle cells (ISCs) | Day 0, Day 15, Day 30, Day 60, Day 90, Day 120.
  Evolution from baseline of the percent of circulating irreversibly sickle cells (ISCs)
Red blood cells (RBC) sickling | Day 0, Day 15, Day 30, Day 60, Day 90, Day 120.
  Evolution from baseline of in vitro Red blood cells (RBC) sickling under hypoxia
Nicotinamide adenine dinucleotide (NAD)+ concentration in whole blood | Day 0, Day 15, Day 30, Day 60, Day 90, Day 120.
  Evolution from baseline of NAD+ concentration in whole blood
β-Nicotinamide mononucleotide (NMN) concentration in whole blood | Day 0, Day 15, Day 30, Day 60, Day 90, Day 120.
  Evolution from baseline of NMN concentration in whole blood
Methyl-Nicotinamide (Me-NAM) concentration in plasma | Day 0, Day 15, Day 30, Day 60, Day 90, Day 120.
  Evolution from baseline of Me-NAM concentration in plasma
Nicotinamide (NAM) concentration in plasma | Day 0, Day 15, Day 30, Day 60, Day 90, Day 120.
  Evolution from baseline of NAM concentration in plasma
Nicotinamide (NAM) concentration in urine | Day 0, Day 15, Day 30, Day 60, Day 90, Day 120.
  Evolution from baseline of NAM concentration in urine
N-Methyl-2-pyridone-5-carboxamide (2PY) concentration in urine | Day 0, Day 15, Day 30, Day 60, Day 90, Day 120.
  Evolution from baseline of 2PY concentration in urine
Change from baseline of self-questionnaire quality of life 36-Item Short Form Survey (SF-36) version 1 | Day 0, Day 15, Day 30, Day 60, Day 90, Day 120.
  Evolutions from baseline in General activity, mood, walking ability, normal work (including housework), relations with other people, sleep, enjoyment of life as measured by the 36-Item Short Form Survey (SF-36) version 1 questionnaire. SF-36 scores range from 0 (worst) to 100 (best)

CONTACTS AND LOCATIONS:
Overall Officials: Laurent LAGANIER, Study Director — LGD SARL; Estelle JEAN-MIGNARD, Principal Investigator — Assistance Publique Hopitaux Marseille
Locations (1):
- Aphm Hopital La Timone Adultes Sce Medecine Interne (Umap), Marseille, France

IPD SHARING:
Plan to Share IPD: No